CLINICAL TRIAL: NCT06393608
Title: If the Use of Epsom Salt (magnesium Sulfate) Compresses 25% Effective in Relieving Perineal Pain in Immediate Postpartum Patients?
Brief Title: Epsom Salt Compresses to Relieve Perineal for Postpartum Care: a Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Antoine Roger (Other)
Collaborators: Hopital Charles Lemoyne (Other); Université de Sherbrooke (Other); Hôpital de Chicoutimi (Unknown); Hôpital Brome-Missisquoi-Perkins (Unknown); Hôpital Honoré-Mercier (Unknown)
Responsible Party: Sponsor-Investigator, Antoine Roger, Dr, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-04-2023-784
Record Dates: First submitted 2024-03-05; First posted 2024-05-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Perineal Injury; Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate; Water

STUDY DESIGN:
Intervention Model Description: The formation of 2 groups will be done randomly. To do this, the Honoré-Mercier Hospital pharmacy will determine the identification of the A and B bottles (containing either the SSE25 or the sterile water) and will communicate it to the other 2 pharmacies. As a result, the pharmacists will be the only ones in the entire study to know the actual contents of each of the A and B bottles. The bottles will be prepared and identified by the pharmacy and given to the mother-child unit of each of the 3 hospitals. Randomization into the two groups will be done in blocks of 6 patients to limit imbalances between the groups. Participants will receive their assigned A or B bottle and the paperwork for postpartum data collection.The randomization group will be recorded on the consent form and data collection documents. Finally, data will be collected to compare the characteristics of the two groups of study participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a triple-blind study. Parturients will be instructed to apply soaked pads (SSE25 or sterile water) for 15 minutes, as needed, four times a day to the perineum, regardless of which group they are in. They will not know the compound in their bottle, they will only know the number of their bottle. The nurses who distribute the bottles to the patients on their shifts will not know which bottle is sterile water and which is SES.25 In addition, each container will be identical and each liquid will have the same texture and color, making it impossible to identify the contents. As described above, the hospital pharmacy will be responsible for preparing bottles and the pharmacy employees will be the only ones who know the contents. Finally, during data analysis, there will be denominationalization of patients and remittance of data that will not be associated with specific intervention groups, so that data analysis will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium sulfate (Active Comparator): Patients in the first group will receive an amber bottle of 250 milliliters containing treatment.The treatment is a solution of MgSO4 25% with sterile water base (Epsom salt solution, concentrated to 25% [SSE25]).
  Interventions: Drug: Epsom salt
- Water (Placebo Comparator): Patients in the second group will receive an amber bottle of 250 milliliters containing the placebo.The placebo is sterile water.
  Interventions: Other: Water

INTERVENTIONS:
Drug: Epsom salt — Epsom salt solution in water, 25% concentration
  Other Names: magnesium sulfate
  Arms: Magnesium sulfate
Other: Water — Water
  Arms: Water

SUMMARY:
The goal of this clinical trial is to determine if topical application of compresses soaked in 25% magnesium sulfate on painful perineum after birth is effective to alleviate pain.

Researchers will compare this treatment to a placebo, compresses soaked in water. Participants will be invited to use their compresses if needed, for 15 minutes, up to four times a day, during their stay at the hospital after giving birth. They will also have to keep a diary of their usage and of their pain.

DETAILED DESCRIPTION:
Background: Despite the high frequency of perineal trauma in obstetrics, management of perineal care and pain is highly variable, relying on very few studies, if any. Treatment of the perineum with compresses soaked in a magnesium sulfate (Epsom salt) solution has not previously been studied but is routinely used in some hospitals in Quebec, Canada. Objectives: This study aims to determine whether compresses soaked in 25% magnesium sulfate in sterile water can alleviate perineal pain in women immediately after childbirth. Population and intervention: Women who have just given birth vaginally and report perineal or vulvar pain of 3/10 or more will be recruited and randomized into an intervention group receiving the treatment (compresses soaked in 25% magnesium sulfate) or a control group receiving a placebo (compresses soaked in water). Methods: This multi-centric, double-blinded randomized clinical trial will be conducted in four hospitals in the province of Quebec, Canada. The investigators plan to recruit a total of 104 participants. Participants will be instructed to apply the compresses on the vulva and perineum for 15 minutes, four times per day, if needed. They will be asked to score their pain before and after using the compresses for the length of their hospital stay, typically between 24 and 48 hours. Secondary outcomes include analgesic use, incidence of complications, participant satisfaction, opinions on feasibility, and any adverse effects caused by the compresses. Discussion: This randomized controlled trial will assess whether the treatment is more effective in relieving pain than the placebo. The study will also determine the safety and feasibility of this method for routine postnatal care. This study could contribute in the long term to the standardization of evidence-based practices for the management of postpartum perineal pain in Canadian hospitals

ELIGIBILITY:
Inclusion Criteria:

* Planned hospital stay at the mother-child unit of the Hôpital de Chicoutimi, Hôpital Charles-Le Moyne, or Hôpital Honoré-Mercier
* Vaginal delivery with or without perineal tear, any degree of tear, including episiotomies
* Obtaining consent for the study
* Languages spoken: French, English or both

Exclusion Criteria:

* Hemodynamic instability
* Surgical procedure such as a cesarean section
* Transfer to another hospital
* Transfer to another care unit
* Chronic use of narcotics
* Inability to complete the logbook
* Unsigned consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Person who has given birth vaginally
Enrollment: 90 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain reduction on the visual and numerical pain scale after each application | 24hours to 48 hours (duration of the stay at the hospital)
  customized visual and numerical pain scale (0-10, 0 being no pain at all and 10 being the worse pain)

SECONDARY OUTCOMES:
other analgesic usage, by filling a medication usage journal | 24hours to 48 hours (duration of the stay at the hospital)
  It includes usually available analgesics, such as acetaminophen, anti-inflammatories, topical analgesics and ice.
Satisfaction, opinions of feasibility through a numerical scale | 24hours to 48 hours (duration of the stay at the hospital)
  Participants will have to fill this part of their diary before they leave the hospital.
Adverse effects, self declared in a journal | 24hours to 48 hours (duration of the stay at the hospital)
  A space in the participant's diary is dedicated for them to declare any benign adverse effects. We don't expect any, since the product is already recognized as safe in literature.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Roger, Principal Investigator — Université de Sherbrooke
Locations (4):
- Canada (4):
  - Hôpital de Chicoutimi, Chicoutimi, Quebec
  - Hôpital Brome-Missisquoi-Perkins, Cowansville, Quebec
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - Hôpital Honoré-Mercier, Saint-Hyacinthe, Quebec